CLINICAL TRIAL: NCT04515719
Title: Efficacy and Safety of Belimumab for Prevention of Disease Flares in SLE Patients With Low Disease Activity
Brief Title: Efficacy and Safety of Belimumab in SLE Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Btrial
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Belimumab; Systemic Lupus Erythematosus; Disease flare
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belimumab 2mg/kg (Experimental): Eligible patients were randomized in a 1:1 ratio to belimumab/placebo on the background of standard therapy. Belimumab 2mg/kg is administered intravenously at week 0, week 2, week 4 and then every 4 weeks until 48 weeks.
  Interventions: Biological: Belimumab
- Placebo (Placebo Comparator): Eligible patients were randomized in a 1:1 ratio to belimumab/placebo on the background of standard therapy. Placebo (normal saline) is administered intravenously at week 0, week 2, week 4 and then every 4 weeks until 48 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Belimumab — Belimumab 2mg/kg intravenously
  Other Names: BENLYSTA™
  Arms: Belimumab 2mg/kg
Biological: Placebo — Placebo intravenously
  Arms: Placebo

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic inflammatory systemic autoimmune disease. Recurrent relapses of disease and development of long-term organ damage are two key unsolved clinical problems. Belimumab is the only FDA-approved biological agent for SLE. Data showed that treatment with belimumab on the background of standard therapy was effective in active SLE patients. However, the efficacy of low-dose belimumab for prevention of disease flares in SLE patients with low disease activity is to be explored.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic systemic autoimmune disease with the incidence of about 70/100,000 in China. Recurrent relapses of disease and development of long-term organ damage are two key unsolved clinical problems. Its pathogenesis is still unclear, but B cells have been confirmed to play a vital role in it. Belimumab, a B-lymphocyte stimulating factor (Blys) inhibitor, was the only FDA-approved biological agent for SLE. BLISS-52 showed that more active lupus patients had their SELENA-SLEDAI score reduced by at least 4 points during 52 weeks with belimumab 10 mg/kg (58% vs 46%, p=0·0024) than with placebo. But there was limited data about belimumab in SLE patients with low disease activity. Our previous study indicated that even these patients still have an annual flare rate of 30-40%. Therefore, we try to explore whether low-dose of belimumab could prevent the disease flares in SLE patients with low disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years;
2. Patients with low disease activity (score≤ 6 at screening on SLEDAI); no British Isles Lupus Assessment Group (BILAG) A and no more than one B;
3. A stable treatment regimen with fixed doses of prednisone (≤ 20mg/day), antimalarial, or immunosuppressive drugs (azathioprine/mycophenolate mofetil/ methotrexate/ciclosporin/leflunomide/tacrolimus) for at least 30 days.
4. Sign the informed consent;

Exclusion Criteria:

1. Alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) > 2 times upper normal limits;
2. Creatinine clearance rate < 60ml/min;
3. Exposure to cyclophosphamide within past 6 months before screening;
4. Exposure to any B cell targeted therapy (Rituximab/belimumab) within past 1 year before screening;
5. History of Malignancy;
6. History of herpes zoster with past 3 months before screening.
7. Chronic HBV/HCV hepatitis；
8. Current infections (HIV/tuberculosis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with disease flares | 52 weeks
  Disease flare is defined by modified SELENA-SLEDAI SLE flare index (SFI).

SECONDARY OUTCOMES:
Percentage of patients with mild/moderate flares | 52 weeks
  Disease flare is defined by modified SELENA-SLEDAI SLE flare index (SFI).
Percentage of patients with major flares | 52 weeks
  Disease flare is defined by modified SELENA-SLEDAI SLE flare index (SFI).
Time to first disease flare | 52 weeks
  Time to first disease flare
prednisone dose at each visit | 52 weeks
  compare the prednisone dose at each visit
SELENA-SLEDAI score at each visit | 52 weeks
  compare the disease activity measured by SELENA-SLEDAI score at each visit
BiLAG score at each visit | 52 weeks
  compare the disease activity measured by BILAG score at each visit
The percentage of patients achieving prednisone-free successfully | 52 weeks
  the percentage of patients achieving prednisone-free successfully
Number of participants with adverse events as assessed by CTCAE v4.0 | 52 weeks
  the safety of belimumab

OTHER OUTCOMES:
Subgroup analysis | 52 weeks
  subgroup analysis aiming to investigate which population will benefit most from belimumab with prespecified factors including age, gender, SLE duration, SELENA- SLEDAI, BILAG, PGA, serology, baseline LLDAS attainment and prednisone dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ye, MD, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Navarra SV, Guzman RM, Gallacher AE, Hall S, Levy RA, Jimenez RE, Li EK, Thomas M, Kim HY, Leon MG, Tanasescu C, Nasonov E, Lan JL, Pineda L, Zhong ZJ, Freimuth W, Petri MA; BLISS-52 Study Group. Efficacy and safety of belimumab in patients with active systemic lupus erythematosus: a randomised, placebo-controlled, phase 3 trial. Lancet. 2011 Feb 26;377(9767):721-31. doi: 10.1016/S0140-6736(10)61354-2. Epub 2011 Feb 4. PMID 21296403
- [Derived] Sun F, Wang H, Zhang D, Shen N, Chen S, Li T, Wan W, Dai SM, Ye S. Low-dose belimumab reduced risk of flares in patients with systemic lupus erythematosus: a multicentre, randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2025 Nov 6:S0003-4967(25)04449-8. doi: 10.1016/j.ard.2025.10.010. Online ahead of print. PMID 41203461
- [Derived] Sun F, Huang W, Chen J, Zhao L, Zhang D, Wang X, Wan W, Dai SM, Chen S, Li T, Ye S. Low-dose belimumab for patients with systemic lupus erythematosus at low disease activity: protocol for a multicentre, randomised, double-blind, placebo-controlled clinical trial. Lupus Sci Med. 2022 Feb;9(1):e000638. doi: 10.1136/lupus-2021-000638. PMID 35105722